CLINICAL TRIAL: NCT01253655
Title: A Phase 1, Open-Label Study To Evaluate 5-HT6 Receptor Occupancy As Measured By Positron Emission Tomography (PET) With Ligand [11C]PF-04171252 Following Single Oral Dose Administration Of PF-05212365 (SAM-531) In Healthy Subjects
Brief Title: To Evaluate The Relationship Between Plasma Drug Levels And Receptor Binding In Brain Using PET (Positron Emission Tomography) In Healthy Volunteers
Acronym: 3193A1-1103
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Yale University (Other)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: B1961009
Record Dates: First submitted 2010-11-02; First posted 2010-12-03 (Estimated); Last update posted 2011-04-28 (Estimated); Status verified 2011-04

CONDITIONS: Healthy
Keywords: Healthy Volunteers
MeSH Terms: interventions — SAM-531

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PF-05212365 (Experimental)
  Interventions: Drug: PF-05212365

INTERVENTIONS:
Drug: PF-05212365 — Single dose of up to 30 mg PF-05212365, delivered as 1 mg, 3 mg, and/or 5 mg on study day 1.
  Other Names: SAM-531

SUMMARY:
The purpose of this study is to evaluate the relationship between plasma drug levels and receptor binding in brain using PET; and to evaluate safety and tolerability after a single administration of PF-05212365 in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects of nonchildbearing potential between the ages of 18 and 55 years, inclusive

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease.
* History of regular alcohol consumption exceeding 7 drinks/week for females or 14 drinks/week for males (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor) within 6 months of screening
* Fulfillment of any of the MRI contraindications on the standard radiography screening questionnaire

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2010-11; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Exposure response of 5-HT6 Receptor Occupancy (RO) of PF-05212365 in the striatum of healthy adult subjects | up to 4 days

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | continuous, up to 4 days
Change from baseline in orthostatic blood pressure | Baseline, -5 pre-dose, and 5, 51, and 72 hrs post-dose
Change from baseline in supine blood pressure | Baseline, -2.5, -1.5, -.5 pre-dose, and 2, 3, 4, 48, 49, 50 hrs post-dose
Change from baseline in Singlet ECG | Baseline and 72 hrs post-dose
Clinically relevant levels of standard hemotology (e.g. Hemoglobin, Hematocrit RBC count), chemistry (e.g. BUN, Creatinine, fasting Glucose), and urinalysis (e.g. pH Glucose, Protein). | Baseline and 72 hrs post-dose
Abnormal findings from standard physical examination | Baseline and 72 hrs post-dose
Maximum concentration (Cmax) for PF-05212365 in plasma | up to 4 days
Time at Cmax (Tmax) for PF-05212365 in plasma | up to 4 days
Area under the concentration-time profile from time zero to the time of the last quantifiableconcentration (AUClast) for PF-05212365 in plasma | up to 4 days
Average concentration during the first post-dose PET scan (Cavg (scan 1)) for PF-05212365 in plasma | 2-4 hrs post-dose
Average concentration during the second post-dose PET scan (Cavg (scan 2)) for PF-05212365 in plasma | 48-50 hrs post dose
Change from baseline in orthostatic pulse rate | Baseline, -5 pre-dose, and 5, 51, and 72 hrs post-dose
Change from baseline in supine pulse rate | Baseline, -2.5, -1.5, -.5 pre-dose, and 2, 3, 4, 48, 49, 50 hrs post-dose
Abnormal findings from standard neurological examination | Baseline and 72 hrs post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1961009&StudyName=To%20Evaluate%20The%20Relationship%20Between%20Plasma%20Drug%20Levels%20And%20Receptor%20Binding%20In%20Brain%20Using%20PET%20%28Positron%20Emission%20Tomography%29%20In%20He